CLINICAL TRIAL: NCT02287493
Title: Pharmacokinetics of Selected Antiinfectives During Sustained Low-efficiency Dialysis (SLED)
Acronym: PhA-SLED
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, PD Dr. rer. medic. Claudia Langebrake, Head Clinical Research Hospital Pharmacy, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: PV4244
Record Dates: First submitted 2014-10-30; First posted 2014-11-10 (Estimated); Results first posted 2021-02-18 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Replacement Therapy, Renal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Meropenem: Adult ICU patients receiving meropenem during SLED will be analyzed for meropenem pharmacokinetics.
  Interventions: Other: Pharmacokinetic Analysis
- Ceftazidim: Adult ICU patients receiving ceftazidim during SLED will be analyzed for ceftazidim pharmacokinetics.
  Interventions: Other: Pharmacokinetic Analysis

INTERVENTIONS:
Other: Pharmacokinetic Analysis

SUMMARY:
In a prospective, non-interventional, monocentric observational study the pharmacokinetic properties of selected antiinfective drugs during sustained low-efficiency dialysis (SLED) will be analyzed.

DETAILED DESCRIPTION:
Antibiotic concentrations are measured whilst patients receive SLED for renal replacement therapy. The plasma specimens will be quantified using high Performance liquid chromatography (HPLC).

Primary endpoint:

- Plasma levels of antiinfectives during SLED

Secondary endpoints:

* mortality
* length of stay at the intensive care unit (ICU) and hospital
* clinical cure of infections

Inclusion criteria:

* age: > 18 years
* patients under SLED
* antiinfective treatment

exclusion criteria:

- missing informed consent

ELIGIBILITY:
Inclusion Criteria:

* age: 18 or older
* patients receiving SLED and either meropenem or ceftazidim

Exclusion Criteria:

* missing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients at University Medical Center Hamburg-Eppendorf receiving SLED and either meropenem or ceftazidim.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kluge, Prof. Dr., Principal Investigator — University Medical Center Hamburg-Eppendorf, Department of Intensive Care
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Braune S, Konig C, Roberts JA, Nierhaus A, Steinmetz O, Baehr M, Kluge S, Langebrake C. Pharmacokinetics of meropenem in septic patients on sustained low-efficiency dialysis: a population pharmacokinetic study. Crit Care. 2018 Jan 30;22(1):25. doi: 10.1186/s13054-018-1940-1. PMID 29382394

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Meropenem | Ceftazidim
Started | 19 | 16
Completed | 19 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Meropenem | Ceftazidim | Total
Number analyzed (Participants) | 19 | 16 | 35
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 66 [52 to 74] | 63 [56 to 67] | 64.5 [33 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 14 | 6 | 20
Region of Enrollment [Number; unit: participants]
  Germany | 19 | 16 | 35

OUTCOME MEASURES:

1. Primary Outcome: Patients Showing Serum Levels of Meropenem or Ceftazidim at the End of SLED Above the Minimal Inhibitory Concentration (MIC)
Description: Plasma concentrations of meropenem or ceftazidim by the end of SLED therapy. Meropenem and ceftazidim are often used for empirical treatment also targeting for Pseudomonas aeruginosa (PSA) infections.
  Therefore, minimal targeted concentrations were set to the MIC of 2 mg/l for meropenem and to the MIC of 4 mg/L for ceftazidime treatment according to the breakpoints of PSA strains.
Time Frame: days receiving SLED, up to 5 days
Measure: Count of Participants; unit: Participants
Groups:
- Meropenem: Adult ICU patients receiving meropenem during SLED will be analyzed for meropenem pharmacokinetics.
  Pharmacokinetic Analysis
- Ceftazidim: Adult ICU patients receiving ceftazidim during SLED will be analyzed for ceftazidim pharmacokinetics.
  Pharmacokinetic Analysis
Arm/Group | Meropenem | Ceftazidim
Number analyzed (Participants) | 19 | 16
Participants
  Trough level < MIC | 0 | 0
  Trough level > MIC | 19 | 16

2. Secondary Outcome: Mortality
Description: ICU mortality
Time Frame: minimum duration of hospital stay, maximum 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Meropenem | Ceftazidim
Number analyzed (Participants) | 19 | 16
Participants | 9 | 9

3. Secondary Outcome: Length of Stay (LOS)
Description: Length of stay at the ICU and in hospital
Time Frame: minimum duration of hospital stay, maximum 1 year
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Meropenem | Ceftazidim
Number analyzed (Participants) | 19 | 16
days
  LOS in hospital | 56 [24 to 264] | 90 [15 to 264]
  LOS in ICU | 36 [8 to 264] | 67 [12 to 264]

4. Secondary Outcome: Number of Patients With Clinical Cure of Infections
Description: Clinical response to antibiotic treatment assessed by laboratory parameters such as leucocyte count, c-reactive protein or procalcitonin levels as well as vasopressor support
Time Frame: minimum duration of hospital stay, maximum 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Meropenem: Adult ICU patients receiving meropenem during SLED will be analyzed
- Ceftazidim: Adult ICU patients receiving ceftazidim during SLED will be analyzed
Arm/Group | Meropenem | Ceftazidim
Number analyzed (Participants) | 19 | 16
Participants | 10 | 9

ADVERSE EVENTS:
Time Frame: Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed. Mortality was not considered to be a Serious Adverse Event.
Description: Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
  Mortality was not considered to be a Serious Adverse Event.
Arm/Group | Meropenem | Ceftazidim
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes